CLINICAL TRIAL: NCT02732691
Title: JENAVALVE ALIGN-AS TRIAL: Safety and Effectiveness/Performance of the Transfemoral JenaValve Pericardial TAVR System in the Treatment of Patients With Symptomatic Severe Aortic Stenosis (AS)
Brief Title: JENAVALVE AS EFS TRIAL: Pericardial TAVR Aortic Stenosis Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: JenaValve Technology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-0003; P02C220_JV06EFS_CIP (Other: JenaValve Technology Inc.); CA-0001 EU (Other: JenaValve Technology Inc.); CA-0001 Germany (Other: JenaValve Technology Inc.); CA-0010 (Other: JenaValve Technology Inc.)
Record Dates: First submitted 2016-03-18; First posted 2016-04-11 (Estimated); Results first posted 2022-11-22 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-10

CONDITIONS: Aortic Valve Stenosis; Heart Valve Diseases; Heart Diseases; Cardiovascular Diseases; Ventricular Outflow Obstruction
Keywords: Valvular Heart Disease; Critical/Severe Aortic Stenosis; High risk symptomatic patients
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Valve Diseases; Heart Diseases; Cardiovascular Diseases; Ventricular Outflow Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transcatheter Aortic Valve Replacement (TAVR) (Experimental): Transcatheter aortic valve replacement (TAVR) will be performed using the JenaValve pericardial valve and delivery system.
  Interventions: Device: JenaValve Pericardial TAVR System

INTERVENTIONS:
Device: JenaValve Pericardial TAVR System — Transcatheter aortic valve replacement (TAVR) will be performed using the JenaValve Pericardial valve and delivery system.

SUMMARY:
To collect information about treatment for severe aortic stenosis (AS), which affects the aortic valve in the heart. Aortic stenosis is a narrowing of the aortic valve opening, which decreases blood flow from the heart and causes symptoms such as chest pain, fainting and shortness of breath. The preferred treatment for severe aortic stenosis is aortic valve replacement surgery.

DETAILED DESCRIPTION:
This study will examine the use of a TAVR (Transcatheter Aortic Valve Replacement), which is a minimally invasive procedure designed to replace the aortic valve inside the heart. This less invasive surgical approach called TAVR is offered to those patients who are high risk for undergoing open heart surgery to replace the aortic valve. In this study, TAVR will be performed using the JenaValve Pericardial TAVR System.

ELIGIBILITY:
Inclusion Criteria:

* Patient with severe degenerative native aortic stenosis (AS).
* Patient at high risk for open surgical valve replacement
* Patient symptomatic according to NYHA functional class II or higher

Exclusion Criteria:

* Congenital uni- or bicuspid aortic valve morphology
* Previous prosthetic aortic valve (bioprosthesis or mechanical) implant
* Endocarditis or other active infection
* Need for urgent or emergent TAVR procedure for any reason
* Cardiogenic shock or hemodynamic instability requiring inotropic support or ventricular assist device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-10-21 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2024-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Martin B Leon, MD, Study Chair — New York-Presbyterian Hospital/Columbia University Medical Center, USA; Torsten P Vahl, MD, Principal Investigator — New York-Presbyterian Hospital/Columbia University Medical Center, USA; Vinod H Thourani, MD, Principal Investigator — Piedmont Heart Institute, USA; Hendrik Treede, MD, Principal Investigator — University Hospital Bonn, Germany
Locations (13):
- United States (2):
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Columbia University Medical Center, New York, New York
- Germany (6):
  - Deutsches Herzzentrum Berlin, Berlin
  - Herzzentrum der Universität zu Köln, Cologne
  - Universitäts-Herzzentrum Freiburg/Bad Krozingen, Freiburg im Breisgau
  - Universitätsklinikum Halle, Halle
  - Universitäres Herzzentrum Hamburg, Hamburg
  - Robert-Bosch-Krankenhaus, Stuttgart
- Netherlands (3):
  - Leiden University Medical Center, Leiden
  - St. Antonius Hospital, Nieuwegein
  - Erasmus University Medical Center, Rotterdam
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Waikato Hospital, Hamilton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zoghbi WA, Adams D, Bonow RO, Enriquez-Sarano M, Foster E, Grayburn PA, Hahn RT, Han Y, Hung J, Lang RM, Little SH, Shah DJ, Shernan S, Thavendiranathan P, Thomas JD, Weissman NJ. Recommendations for Noninvasive Evaluation of Native Valvular Regurgitation: A Report from the American Society of Echocardiography Developed in Collaboration with the Society for Cardiovascular Magnetic Resonance. J Am Soc Echocardiogr. 2017 Apr;30(4):303-371. doi: 10.1016/j.echo.2017.01.007. Epub 2017 Mar 14. No abstract available. PMID 28314623
- [Background] Nishimura RA, Otto CM, Bonow RO, Carabello BA, Erwin JP 3rd, Fleisher LA, Jneid H, Mack MJ, McLeod CJ, O'Gara PT, Rigolin VH, Sundt TM 3rd, Thompson A. 2017 AHA/ACC Focused Update of the 2014 AHA/ACC Guideline for the Management of Patients With Valvular Heart Disease: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Circulation. 2017 Jun 20;135(25):e1159-e1195. doi: 10.1161/CIR.0000000000000503. Epub 2017 Mar 15. No abstract available. PMID 28298458
- [Background] Iung B, Baron G, Butchart EG, Delahaye F, Gohlke-Barwolf C, Levang OW, Tornos P, Vanoverschelde JL, Vermeer F, Boersma E, Ravaud P, Vahanian A. A prospective survey of patients with valvular heart disease in Europe: The Euro Heart Survey on Valvular Heart Disease. Eur Heart J. 2003 Jul;24(13):1231-43. doi: 10.1016/s0195-668x(03)00201-x. PMID 12831818
- [Background] Hamid N, Ranard LS, Khalique OK, Hahn RT, Nazif TM, George I, Ng V, Leon MB, Kodali SK, Vahl TP. Commissural Alignment After Transfemoral Transcatheter Aortic Valve Replacement With the JenaValve Trilogy System. JACC Cardiovasc Interv. 2021 Sep 27;14(18):2079-2081. doi: 10.1016/j.jcin.2021.07.025. No abstract available. PMID 34556282

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Transcatheter Aortic Valve Replacement (TAVR)
Started | 68
Completed | 68
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Enrolled
Arm/Group | Transcatheter Aortic Valve Replacement (TAVR)
Number analyzed (Participants) | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 83 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: All-Cause Mortality
Description: All-cause mortality rate at 30 Day
Time Frame: 30 Day
Population: Enrolled
Measure: Count of Participants; unit: Participants
Arm/Group | Transcatheter Aortic Valve Replacement (TAVR)
Number analyzed (Participants) | 68
Participants | 2

2. Secondary Outcome: Myocardial Infarction
Description: Peri-procedural and spontaneous myocardial infarction
Time Frame: 30 Day
Measure: Count of Participants; unit: Participants
Arm/Group | Transcatheter Aortic Valve Replacement (TAVR)
Number analyzed (Participants) | 68
Participants | 1

3. Secondary Outcome: All Stroke/TIA
Description: Neurological Complications
Time Frame: 30 Day
Measure: Count of Participants; unit: Participants
Arm/Group | Transcatheter Aortic Valve Replacement (TAVR)
Number analyzed (Participants) | 68
Participants | 6

4. Secondary Outcome: Major Bleeding
Description: Life threatening or major bleeding
Time Frame: 30 Day
Measure: Count of Participants; unit: Participants
Arm/Group | Transcatheter Aortic Valve Replacement (TAVR)
Number analyzed (Participants) | 68
Participants | 4

5. Secondary Outcome: Major Vascular Complication
Description: Major vascular and bleeding complications
Time Frame: 30 Day
Measure: Count of Participants; unit: Participants
Arm/Group | Transcatheter Aortic Valve Replacement (TAVR)
Number analyzed (Participants) | 68
Participants | 5

6. Secondary Outcome: Conduction Disturbance and Arrhythmias
Description: Conduction system injury (defect), including AV block, which may require a permanent pacemaker
Time Frame: 30 Day
Measure: Count of Participants; unit: Participants
Arm/Group | Transcatheter Aortic Valve Replacement (TAVR)
Number analyzed (Participants) | 68
Participants | 10

7. Secondary Outcome: Acute Kidney Injury (AKI)
Description: Number of patients who were diagnosed with AKI Stage 2 or 3:
  AKI Stage 2: Increase in serum creatinine to 200%-299% (2.0%-2.99% increase compared with baseline) OR urine output <0.5 mL/kg/h for >12 but <24 h
  AKI Stage 3: Increase in serum creatinine to ≥300% (>3 × increase compared with baseline) OR serum creatinine of ≥4.0 mg/dL (≥354 mmol/L) with an acute increase of at least 0.5 mg/dL (44 mmol/L) OR urine output <0.3 ml/kg/h for ≥24 h OR anuria for ≥12 h
Time Frame: 30 Day
Measure: Count of Participants; unit: Participants
Arm/Group | Transcatheter Aortic Valve Replacement (TAVR)
Number analyzed (Participants) | 68
Participants | 0

8. Secondary Outcome: Coronary Obstruction Requiring Intervention
Description: Coronary obstruction post-implant requiring intervention
Time Frame: 30 Day
Measure: Count of Participants; unit: Participants
Arm/Group | Transcatheter Aortic Valve Replacement (TAVR)
Number analyzed (Participants) | 68
Participants | 0

9. Secondary Outcome: Endocarditis
Description: Bacterial endocarditis
Time Frame: 30 Day
Measure: Count of Participants; unit: Participants
Arm/Group | Transcatheter Aortic Valve Replacement (TAVR)
Number analyzed (Participants) | 68
Participants | 0

10. Secondary Outcome: Conversion to Surgical Aortic Valve Replacement (SAVR)
Description: Number of patients who underwent conversion to open sternotomy during the TAVR procedure secondary to any procedure-related complications
Time Frame: 30 Day
Measure: Count of Participants; unit: Participants
Arm/Group | Transcatheter Aortic Valve Replacement (TAVR)
Number analyzed (Participants) | 68
Participants | 1

11. Secondary Outcome: THV Malpositioning
Description: Number of patients who experienced:
  Migration: After initial correct positioning, the valve prosthesis moves upwards or downwards, within the aortic annulus from its initial position, with or without consequences
  Embolization: The valve prosthesis moves during or after deployment such that it loses contact with the aortic annulus
  Ectopic Valve Deployment: Permanent deployment of the valve prosthesis in a location other than the aortic root
Time Frame: 30 Day
Measure: Count of Participants; unit: Participants
Arm/Group | Transcatheter Aortic Valve Replacement (TAVR)
Number analyzed (Participants) | 68
Participants | 3

ADVERSE EVENTS:
Time Frame: 30 day
Arm/Group | Transcatheter Aortic Valve Replacement (TAVR)
All-Cause Mortality (participants affected / at risk) | 2/68
Serious Adverse Events (participants affected / at risk) | 39/68
Other Adverse Events (participants affected / at risk) | 23/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Transcatheter Aortic Valve Replacement (TAVR) (N=68)
Access Site Disection (Injury, poisoning and procedural complications) | 1
Acute Coronary Syndrome (Cardiac disorders) | 1
Acute Pancreatitis Secondary To Retained Gallstones (Hepatobiliary disorders) | 1
Allergic Reaction (General disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Aortic Rupture (Cardiac disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Arterial Occlusion (Cardiac disorders) | 2
Arterial Occlusive Desease (Cardiac disorders) | 1
Bilious Attack (Hepatobiliary disorders) | 1
Bleeding (Life Threatening/Disabling) (Blood and lymphatic system disorders) | 1
Bleeding (Major) (Blood and lymphatic system disorders) | 3
Bleeding Complication (Blood and lymphatic system disorders) | 5
Bradycardia (Cardiac disorders) | 1
Cellulitus (Infections and infestations) | 1
Cerebral Hypoxia Due To Open Heart Surgery. Therefore Cerebral Iscemia Which Was Leading To Death. (Nervous system disorders) | 1
Conduction Disturbance (Cardiac disorders) | 5
Deep Vein Thrombosis (Vascular disorders) | 1
Ectopic Deployment (Injury, poisoning and procedural complications) | 1
Exacerbation COPD (Respiratory, thoracic and mediastinal disorders) | 2
Exacerbation Of COPD (Respiratory, thoracic and mediastinal disorders) | 1
Fall Secondary To Postural Hypotension (General disorders) | 1
Febrile But No Infection Identified (General disorders) | 1
Fluid Overload Secondary To Fludricortisone Use (General disorders) | 1
Gastroenteritis (Gastrointestinal disorders) | 1
Gastroenteritis Norovirus (Gastrointestinal disorders) | 1
GI Complication (Gastrointestinal disorders) | 3
Heart Failure (Cardiac disorders) | 3
Hematoma (Injury, poisoning and procedural complications) | 1
Hypertension (Vascular disorders) | 2
Infection/Inflammation (Infections and infestations) | 1
INR > 8 And General Weakness (General disorders) | 1
Maxillary Fracture (Le-Fort I Fracture) (General disorders) | 1
Medication Reaction (General disorders) | 1
Multiple Falls Secondary To Medication And Parkinsons (General disorders) | 1
Myocardial Insufficiency (Cardiac disorders) | 1
Neurological Event (Nervous system disorders) | 1
Other Infection (Infections and infestations) | 8
Pancolitis (Gastrointestinal disorders) | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonia (Infections and infestations) | 3
Premature Valve Deployment (Injury, poisoning and procedural complications) | 1
Pseudomonas Bacteremia (Infections and infestations) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Recurring Subdural Hematoma (Injury, poisoning and procedural complications) | 1
Reduced Mobility (General disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Restenosis (Cardiac disorders) | 1
Sepsis (Infections and infestations) | 1
Spondylolisthesis/Foraminal Stenosis (Musculoskeletal and connective tissue disorders) | 1
Status Epilepticus (Nervous system disorders) | 1
Stroke/TIA (Nervous system disorders) | 4
Subacute Cerebal Infarct Bilaterally. (Nervous system disorders) | 1
Subdural Hematoma (Injury, poisoning and procedural complications) | 1
Suspected Endocarditis (Infections and infestations) | 1
Syncope (Nervous system disorders) | 1
Tooth Extraction (General disorders) | 1
Urosepsis (Infections and infestations) | 1
Valve Malposition / Ectopic Deployment (Injury, poisoning and procedural complications) | 1
Vascular Dissection (Vascular disorders) | 1
Worsening Of Atrial Fibrilation (Cardiac disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Transcatheter Aortic Valve Replacement (TAVR) (N=68)
Bleeding Complication (Blood and lymphatic system disorders) | 5
Chest Pain (General disorders) | 4
Other (General disorders) | 17
Respiratory Complication (Respiratory, thoracic and mediastinal disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-15): https://cdn.clinicaltrials.gov/large-docs/91/NCT02732691/Prot_SAP_000.pdf